CLINICAL TRIAL: NCT05873374
Title: A Phase 2 Study to Evaluate the Safety, Tolerability, Reactogenicity, and Immunogenicity of Baiya SARS-CoV-2 Vax 2 Vaccine as a Booster Following Vaccination for COVID-19 in Adults Between 18 and 64 Years
Brief Title: Evaluation of Safety, Tolerability, Reactogenicity, Immunogenicity of Baiya SARS-CoV-2 Vax 2 as a Booster for COVID-19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Baiya Phytopharm Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Baiya-Vax2-P2a-Boost
Record Dates: First submitted 2023-05-23; First posted 2023-05-24 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: COVID-19 Vaccine; COVID-19
Keywords: SARS-CoV-2; SARS-CoV-2 vaccine; COVID-19; COVID-19 Vaccine; Booster vaccine; Plant vaccine
MeSH Terms: conditions — COVID-19 | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The treatment will be masked to the participants and site staff (including the investigators and the care providers which are blinded site staff).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 50 μg Baiya SARS-CoV-2 Vax 2 (Experimental): 0.5 mL of Baiya SARS-CoV-2 Vax 2 Vaccine as a booster dose via IM injection on Day 1 for adult participants (18 - 64 years old)
  Interventions: Biological: 50 μg Baiya SARS-CoV-2 Vax 2
- Placebo (Placebo Comparator): 0.5 mL of placebo via IM injection on Day 1 for adult participants (18 - 64 years old)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: 50 μg Baiya SARS-CoV-2 Vax 2 — Intramuscular injection in the deltoid region of 0.5 mL/dose of 50 μg Baiya SARS-CoV-2 Vax 2
  Arms: 50 μg Baiya SARS-CoV-2 Vax 2
Other: Placebo — Intramuscular injection in the deltoid region of 0.5 mL/dose of 0.9% Sodium Chloride
  Other Names: 0.9% Sodium Chloride
  Arms: Placebo

SUMMARY:
The investigational product Baiya SARS-CoV-2 Vax 2 vaccine is a second-generation of protein subunit vaccine from plant to prevent COVID-19 disease.

This is a Phase 2, randomised, and double-blinded study to assess the safety, tolerability, reactogenicity and immunogenicity of Baiya SARS-CoV-2 Vax 2 vaccine, when used as a booster vaccination following vaccination with the alternate and widely used COVID-19 vaccines.

DETAILED DESCRIPTION:
This is a Phase 2, randomised, and double-blinded study. The participants will be randomised to receive either the investigational product or the placebo at a ratio of 2:1. 0.5 mL of the assigned vaccine will be administered as an IM injection. Each participant will be followed up for 6 months after vaccination.

The primary objective aims to assess the safety, tolerability, and reactogenicity of Baiya SARS-CoV-2 Vax 2 vaccine in adults (18-64 years old) as a booster vaccination following vaccination with the alternate and widely used COVID-19 vaccines.

The secondary objective aims to evaluate safety, tolerability, reactogenicity, and immunogenicity up to 28 days after the booster vaccination.

An interim analysis of all safety and available immunogenicity data up to Visit 6 (Day 29 ±3) will be conducted for the DSMB review.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol
2. Participant must be able to comply with study procedures and be available for all study visits.
3. Previously receive COVID-19 vaccines either homologous or heterologous vaccination at least 3 doses and the last booster dose for more than 6 months prior to Visit 2 (Day 1).
4. Be aged between 18 and 64 years, inclusive, at the time of signing informed consent
5. Have a BMI between 18.5 and 35.0 kg/m2 inclusive
6. Healthy as determined by the Investigator based on pre-study medical history, physical examination and vital signs
7. Males must be surgically sterile (> 30 days since vasectomy with no viable sperm), practice true abstinence, or, if engaged in sexual activities with a female with childbearing potential, use condoms from the time of vaccination until 60 days after the vaccination
8. Females of childbearing potential must practice true abstinence, or, if engaged in sexual activities with a male, agree to use highly effective (failure rate of <1% per year when used consistently and correctly), double-barrier contraceptive measures* for at least 60 days following vaccination.

   * PI to assess the suitability of contraceptive measures on a case-by-case basis. The measures can include: combined (estrogen and progestogen) hormonal contraception associated with inhibition of ovulation, progestogen-only hormonal contraception associated with inhibition of ovulation, intrauterine device, intrauterine hormone releasing system, and documented bilateral tubal occlusion hysterectomy, bilateral salpingectomy, bilateral Essure® placement, and bilateral ovariectomy.

Exclusion Criteria:

1. Known history of COVID-19 infection within 6 months at screening or Visit 2 (Day 1).

   Participants who screen-fail on this criterion may be rescreened.
2. Have received any investigational COVID-19 vaccine.
3. Have received any other vaccine within 30 days prior to Visit 2 (Day 1) or plan to receive any other vaccine within 30 days after Visit 2 (Day 1) as per the investigator's judgment. Participants who screen-fail on this criterion may be rescreened.
4. Have an ongoing AE assessed as related to any prior COVID-19 vaccine or COVID-19 disease as per the investigator's judgment.
5. Women who are pregnant, breast feeding or planning to become pregnant within 60 days of vaccination and men who plan to conceive a child within 60 days of vaccination.
6. Has a clinically unstable chronic underlying disease such as hypertension, diabetes mellitus, chronic obstructive pulmonary disease, asthma, or any other condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant or that could prevent, confound, or limit the assessments specified in the protocol.

   Except for stable symptoms and signs that are medically controlled in the judgment of the investigator, which can be enrolled.
7. Anticipating the need for immunosuppressive treatment within the 6 months following Visit 2 (Day 1).
8. Being treated with other registered or investigational drug for prophylaxis or treatment of COVID-19 such as EVUSHELD or receive within 6 months prior to vaccination or plan to receive within 6 months after vaccination.
9. Immunosuppressive illness or immunodeficient state, including hematologic malignancy, history of solid organ or bone marrow transplantation, asplenia, primary immunodeficiency diseases and HIV infection.
10. Cancer or any malignancy that has been in remission for less than 5 years, except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
11. Administration of other investigational products, or blood products within 4 weeks prior to Visit 2 (Day 1) or planned administration of investigational products, blood products, blood or tissue donation, or blood transfusion within 6 months after Visit 2 (Day 1).
12. Clinically significant abnormalities in clinical laboratory tests during Screening in the opinion of the Investigator.
13. Presence of self-reported or medically documented significant medical or psychiatric condition(s) that as judged by the investigator(s) may not be in the participants' interest to participate in the study.
14. History of severe allergy (requiring hospital care), anaphylaxis, severe reaction to any drug or prior vaccination, or any known or suspected allergies or sensitivities to any component of the investigational vaccine or tobacco.
15. History of systemic steroids (prednisone ≥ 20 mg/day for >14 consecutive days) within 3 months prior to screening. Topical, inhaled, intranasal, and intra-articular corticosteroids are allowed regardless of dose.
16. Receipt of immunoglobulins or blood products within 90 days prior to vaccination or planned treatment during the study periods.
17. Thrombocytopenia or other coagulation disorders for whom IM injections are contraindicated or receiving anticoagulant therapy.*

    * Anticoagulant therapy: continuous use of anticoagulants such as coumarin/warfarin or new oral anticoagulants/antiplatelets. The use of aspirin or clopidogrel is acceptable.
18. Alcoholism, history of alcohol or drug abuse that, in the opinion of the PI, could affect the participant's safety or compliance with study, or chronic liver disease such as cirrhosis at screening.
19. Have received any investigational drug from 30 days prior to Screening until 30 days after receiving the assigned vaccination in this study.
20. The Investigator, sub-Investigator, study staff, sponsor, pharmaceutical product development or their family members.
21. Presence of tattoo, bruising, or other skin blemish at the administration site that would, in the opinion of the Investigator, inhibit the ability to perform an assessment of local tolerability.
22. Positive HBsAg, anti-HCV or anti-HIV tests at Screening
23. Active COVID-19 infection or COVID-19 positive based on ATK testing at screening or Visit 2 (Day 1).
24. Presence of an acute illness, as determined by the Investigator(s), with or without fever (forehead temperature measured with validated device ≥ 37.5oC) within 72 hours prior to vaccination. Participants who screen-fail on this criterion may be rescreened following a suitable recovery period as determined by the Investigator(s).
25. Receipt of herbal medicine (such as products of Andrographis paniculata) within 5 days prior to vaccine administration or within 6 months after vaccination.
26. Any other reason which, in the opinion of the Investigator, makes the individual ineligible for the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Number, percentage, and severity of solicited local and systemic reactogenicity AEs | 7-day post administration
Number, percentage, and severity of unsolicited AEs | Day 1 to 28 days after administration
Number, percentage, and severity of treatment-related AEs | Day 1 to 28 days after administration
Abnormal clinically significant changes in clinical laboratory tests (haematology, coagulation, chemistry, and urinalysis) | Day 1 to 28 days after administration
Abnormal clinically significant changes in vital signs | Day 1 to 28 days after administration
Abnormal clinically significant physical examination | Day 1 to 28 days after administration

SECONDARY OUTCOMES:
Geometric Mean Titres (GMT) of SARS-CoV-2 specific serum neutralizing antibody (MicroVNT) | at 7, 14, 21 and 28 days after administration
Geometric Mean Fold Rises (GMFR) of SARS-CoV-2 specific serum neutralizing antibody (MicroVNT) | at 7, 14, 21 and 28 days after administration
Seroconversion Rate of SARS-CoV-2 specific serum neutralizing antibody (MicroVNT) | at 7, 14, 21 and 28 days after administration
  Seroconversion Rate is defined as the proportion of participants who achieves a greater than or equal to 4-fold rise from baseline
GMT of SARS-CoV-2-surrogate viral neutralising antibody | at 7, 14, 21 and 28 days after administration
  measured by surrogate antibody ELISA
GMFR of SARS-CoV-2-surrogate viral neutralising antibody | at 7, 14, 21 and 28 days after administration
  measured by surrogate antibody ELISA
Seroconversion Rate of SARS-CoV-2-surrogate viral neutralising antibody | at 7, 14, 21 and 28 days after administration
  measured by surrogate antibody ELISA
GMT of SARS-CoV-2 variants pseudovirus-specific serum neutralising antibody | at 14 and 28 days after administration
GMFR of SARS-CoV-2 variants pseudovirus-specific serum neutralising antibody | at 14 and 28 days after administration
Seroconversion Rate of SARS-CoV-2 variants pseudovirus-specific serum neutralising antibody | at 14 and 28 days after administration
GMT of SARS-CoV-2 RBD-specific IgG antibody | at 7, 14, 21 and 28 days after administration
  measured by ELISA
GMFR of SARS-CoV-2 RBD-specific IgG antibody | at 7, 14, 21 and 28 days after administration
  measured by ELISA
Seroconversion Rate of SARS-CoV-2 RBD-specific IgG antibody | at 7, 14, 21 and 28 days after administration
  measured by ELISA
Percentage of participants who have positive specific CD4 and CD8 T-cell IFNγ ELISpot responses (detectable above the assay cut-off) | at 7, 14, 21 and 28 days after administration
  SARS-CoV-2 RBD-specific CD4+ and CD8+ T-cell responses as measured by IFNγ ELISpot assay
Median number of spot-forming cells (SFC) per 1 million PBMCs | at 7, 14, 21 and 28 days after administration
  SARS-CoV-2 RBD-specific CD4+ and CD8+ T-cell responses as measured by IFNγ ELISpot assay
Percentage of participants who show positive specific Th1 responses, or Th2 responses (detectable above the assay cut-off) | at 7, 14, 21 and 28 days after administration
  SARS-CoV-2 RBD-specific Th1/Th2 polarisation responses quantified by intracellular cytokine staining
Median percentage specific Th1/Th2 response of each cohort | at 7, 14, 21 and 28 days after administration
  SARS-CoV-2 RBD-specific Th1/Th2 polarisation responses quantified by intracellular cytokine staining
Number and percentage of serious adverse events (SAEs) | up to 6 months after administration

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Saovabha Memorial Institute, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No